CLINICAL TRIAL: NCT00996606
Title: Open Label, Multicentric Phase IIIb Study to Evaluate the Effect of Tocilizumab in Combination With DMARDs in the Inhibition of Progression of Synovitis, Bone Marrow Edema, and Erosions Evaluated by Dedicated Magnetic Resonance Imaging (MRI) in the Hand of Patients With Rheumatoid Arthritis (RA)
Brief Title: A Study of Tocilizumab in Combination With Disease-Modifying Anti-Rheumatic Drugs (DMARDs) in Participants With Moderate to Severe Active Rheumatoid Arthritis With an Inadequate Response to DMARDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22413; 2009-012185-32
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents; tocilizumab

ARMS (1):
- Tocilizumab in Active RA (Experimental): Participants with active RA will receive tocilizumab as 8 mg/kg via IV infusion every 4 weeks. A total of 12 infusions will be given from Baseline to Week 44, and participants will be assessed through Week 48.
  Interventions: Drug: DMARDs; Drug: Tocilizumab

INTERVENTIONS:
Drug: DMARDs — Participants may continue on a stable dose of their current DMARD therapy as prescribed. The choice of DMARD is at the discretion of the treating physician and is not specified by the protocol.
Drug: Tocilizumab — Tocilizumab will be given as 8 mg/kg via IV infusion every 4 weeks for a total of 12 infusions. The maximum allowed dose is 800 mg.
  Other Names: RoActemra, Actemra

SUMMARY:
This open-label, single-arm study will evaluate the efficacy and safety of tocilizumab in combination with DMARDs in participants with moderate to severe active rheumatoid arthritis who have an inadequate response to DMARDs. Participants will receive tocilizumab as 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion every 4 weeks in addition to their current DMARD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active RA of ≥6 months duration
* DAS28 >3.2
* Inadequate response to a stable dose of non-biologic DMARD for ≥2 months
* Those receiving oral corticosteroids must have been at stable dose for ≥25 days in the 28 days prior to first study treatment

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA
* History of or current inflammatory joint disease other than RA
* Previous treatment with alkylating agents or total lymphoid irradiation
* Intra-articular or parenteral corticosteroids within 6 weeks prior to Baseline
* Previous treatment with any cell-depleting therapies
* American College of Rheumatology (ACR) Functional Class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Italy (10):
  - Coppito, Abruzzo
  - Napoli, Campania
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Pavia, Lombardy
  - Palermo, Sicily
  - Pisa, Tuscany
  - Cona (Ferrara), Veneto
  - Padua, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab in Active Rheumatoid Arthritis (RA): Participants with active RA received tocilizumab as 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion every 4 weeks. A total of 12 infusions were given from Baseline to Week 44, and participants were assessed through Week 48.
Period: Overall Study
Arm/Group | Tocilizumab in Active Rheumatoid Arthritis (RA)
Started | 58
Completed | 50
Not Completed | 8
Not completed — Adverse Event or Intercurrent Illness | 2
Not completed — Insufficient Therapeutic Response | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of study medication.
Groups:
- Tocilizumab in Active RA: Participants with active RA received tocilizumab as 8 mg/kg via IV infusion every 4 weeks. A total of 12 infusions were given from Baseline to Week 44, and participants were assessed through Week 48.
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Synovitis of the Wrist According to Rheumatoid Arthritis Magnetic Resonance Imaging (RAMRIS) Score
Description: Synovitis of the wrist was assessed at three sites including the radioulnar joint (RUJ), the radiocarpal joint (RCJ), and the intercarpal-carpometacarpal joints (IC-CMCJ). Global RAMRIS scores were assigned on a scale of 0 to 3 at each site, where 0 represented normal appearance with no synovial enhancement and each 1-point increase reflected one-third of the presumed maximum volume of enhancing tissue in the synovial compartment. The scores for all three sites were added to give an aggregated score of 0 to 9. Baseline absolute value (AV) and change from Baseline to Week 4 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Week 4
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who contributed to the endpoint. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 55
units on a scale
  Baseline AV (n=55) | 5.78 (2.72)
  Week 4 (n=49) | -0.88 (1.56)

2. Primary Outcome: Change From Baseline to Week 4 in Synovitis of the Wrist According to Relative Enhancement (RE) Before and After Contrast Injection
Description: RE was calculated as [S0 minus (-) S55] divided by (÷) S0, multiplied by (×) 100 percent (%), where S0 was defined as the signal noise ratio before contrast injection, and S55 was defined as the signal noise ratio 55 seconds after injection. Signal noise ratios were measured as the ratio between the signal in the region of interest and the standard deviation of background noise. Baseline AV and change from Baseline to Week 4 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent relative enhancement
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 54
percent relative enhancement
  Baseline AV (n=54) | 99.25 (57.85)
  Week 4 (n=45) | -0.48 (47.85)

3. Primary Outcome: Change From Baseline to Week 4 in Synovitis of the Wrist According to Rate of Early Enhancement (REE) Per Second Before and After Contrast Injection
Description: REE per second was calculated as [S55 - S0] ÷ [S0 × 55 seconds] × 100%, where S0 was defined as the signal noise ratio before contrast injection, and S55 was defined as the signal noise ratio 55 seconds after injection. Signal noise ratios were measured as the ratio between the signal in the region of interest and the standard deviation of background noise. Baseline AV and change from Baseline to Week 4 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent rate of early enhancement
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 54
percent rate of early enhancement
  Baseline AV (n=54) | 1.19 (1.04)
  Week 4 (n=45) | -0.10 (0.86)

4. Secondary Outcome: Change From Baseline to Weeks 2, 12, 24, and 48 in Synovitis of the Wrist According to RAMRIS Score
Description: Synovitis of the wrist was assessed at three sites including the RUJ, the RCJ, and the IC-CMCJ. Global RAMRIS scores were assigned on a scale of 0 to 3 at each site, where 0 represented normal appearance with no synovial enhancement and each 1-point increase reflected one-third of the presumed maximum volume of enhancing tissue in the synovial compartment. The scores for all three sites were added to give an aggregated score of 0 to 9. The changes from Baseline to Weeks 2, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Weeks 2, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 50
units on a scale
  Week 2 (n=45) | -0.44 (1.03)
  Week 12 (n=50) | -1.28 (1.96)
  Week 24 (n=49) | -1.94 (2.34)
  Week 48 (n=47) | -1.60 (2.42)

5. Secondary Outcome: Change From Baseline to Weeks 2, 12, 24, and 48 in Synovitis of the Wrist According to RE Before and After Contrast Injection
Description: RE was calculated as [S0 - S55] ÷ S0 × 100%, where S0 was defined as the signal noise ratio before contrast injection, and S55 was defined as the signal noise ratio 55 seconds after injection. Signal noise ratios were measured as the ratio between the signal in the region of interest and the standard deviation of background noise. The changes from Baseline to Weeks 2, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Weeks 2, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent relative enhancement
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percent relative enhancement
  Week 2 (n=44) | 5.80 (46.14)
  Week 12 (n=49) | -9.27 (50.07)
  Week 24 (n=48) | -26.48 (57.99)
  Week 48 (n=45) | -19.74 (74.08)

6. Secondary Outcome: Change From Baseline to Weeks 2, 12, 24, and 48 in Synovitis of the Wrist According to REE Per Second Before and After Contrast Injection
Description: REE per second was calculated as [S55 - S0] ÷ [S0 × 55 seconds] × 100%, where S0 was defined as the signal noise ratio before contrast injection, and S55 was defined as the signal noise ratio 55 seconds after injection. Signal noise ratios were measured as the ratio between the signal in the region of interest and the standard deviation of background noise. The changes from Baseline to Weeks 2, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Weeks 2, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent rate of early enhancement
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percent rate of early enhancement
  Week 2 (n=44) | -0.04 (1.11)
  Week 12 (n=49) | -0.48 (0.96)
  Week 24 (n=48) | -0.57 (0.87)
  Week 48 (n=45) | -0.66 (1.24)

7. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Synovitis of the Wrist and Metacarpo-Phalangeal (MCP) Joints According to Modified RAMRIS Score
Description: Synovitis of the wrist was assessed at three sites including the RUJ, the RCJ, and the IC-CMCJ. Global RAMRIS scores were assigned on a scale of 0 to 3 at each site, where 0 represented normal appearance with no synovial enhancement and each 1-point increase reflected one-third of the presumed maximum volume of enhancing tissue in the synovial compartment. The scores for all three sites were added to give an aggregated score of 0 to 9. Synovitis of MCP joints was determined on the basis of Short Inversion Time Inversion Recovery (STIR) sequence evaluation with modification of the RAMRIS score. Four MCP joint compartments were each assessed 0 to 3, so the aggregated MCP joint score ranged from 0 to 12. Combined synovitis in wrist and MCP joints was determined on the basis of STIR sequences to produce overall score from 0 to 21. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, 48 were averaged among all participants, where negative changes indicated improvement in synovitis.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 55
units on a scale
  Wrist Global Score, Baseline AV (n=55) | 5.04 (2.24)
  Wrist Global Score, Week 2 (n=45) | -0.02 (1.70)
  Wrist Global Score, Week 4 (n=50) | -0.20 (1.50)
  Wrist Global Score, Week 12 (n=51) | -0.47 (2.07)
  Wrist Global Score, Week 24 (n=50) | -1.06 (2.11)
  Wrist Global Score, Week 48 (n=47) | -1.23 (2.28)
  Wrist Distal RUJ Score, Baseline AV (n=53) | 1.62 (0.95)
  Wrist Distal RUJ Score, Week 2 (n=43) | -0.09 (0.78)
  Wrist Distal RUJ Score, Week 4 (n=48) | -0.15 (0.62)
  Wrist Distal RUJ Score, Week 12 (n=48) | -0.21 (0.87)
  Wrist Distal RUJ Score, Week 24 (n=48) | -0.44 (0.74)
  Wrist Distal RUJ Score, Week 48 (n=45) | -0.58 (0.94)
  Wrist Distal RCJ Score, Baseline AV (n=55) | 1.73 (0.78)
  Wrist Distal RCJ Score, Week 2 (n=45) | 0.11 (0.80)
  Wrist Distal RCJ Score, Week 4 (n=50) | -0.06 (0.62)
  Wrist Distal RCJ Score, Week 12 (n=51) | -0.12 (0.77)
  Wrist Distal RCJ Score, Week 24 (n=50) | -0.30 (0.91)
  Wrist Distal RCJ Score, Week 48 (n=47) | -0.38 (0.92)
  Wrist IC-CMCJ Score, Baseline AV (n=55) | 1.75 (0.89)
  Wrist IC-CMCJ Score, Week 2 (n=44) | 0.00 (0.72)
  Wrist IC-CMCJ Score, Week 4 (n=50) | 0.00 (0.70)
  Wrist IC-CMCJ Score, Week 12 (n=51) | -0.22 (0.88)
  Wrist IC-CMCJ Score, Week 24 (n=50) | -0.40 (0.88)
  Wrist IC-CMCJ Score, Week 48 (n=47) | -0.34 (0.96)
  MCP STIR Joint Score, Baseline AV (n=54) | 4.57 (3.10)
  MCP STIR Joint Score, Week 2 (n=40) | -0.13 (1.76)
  MCP STIR Joint Score, Week 4 (n=47) | -0.53 (1.90)
  MCP STIR Joint Score, Week 12 (n=45) | -0.53 (2.07)
  MCP STIR Joint Score, Week 24 (n=46) | -1.02 (2.24)
  MCP STIR Joint Score, Week 48 (n=44) | -1.25 (2.53)
  Wrist and MCP Aggregate Score, Baseline AV (n=56) | 9.36 (4.49)
  Wrist and MCP Aggregate Score, Week 2 (n=46) | -0.54 (2.67)
  Wrist and MCP Aggregate Score, Week 4 (n=50) | -0.74 (2.62)
  Wrist and MCP Aggregate Score, Week 12 (n=51) | -1.33 (3.58)
  Wrist and MCP Aggregate Score, Week 24 (n=50) | -2.24 (3.54)
  Wrist and MCP Aggregate Score, Week 48 (n=47) | -2.49 (3.59)

8. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Number of Bones With Erosion in the Wrist and MCP Joints
Description: Erosion was evaluated at 15 sites in the wrist and 8 sites in the MCP joints. Bone erosion was scored on a scale of 0 to 10, where 0 represented no bone erosion and each 1-point increase reflected up to a 10% increase in extent of erosion. The number of bones with erosion was taken as the count of joints with a bone erosion score greater than or equal to (≥) 1. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in erosion.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bones with erosion
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
bones with erosion
  Baseline AV (n=56) | 8.07 (4.71)
  Week 2 (n=46) | -0.26 (1.16)
  Week 4 (n=50) | -0.16 (1.04)
  Week 12 (n=51) | -0.14 (1.61)
  Week 24 (n=50) | -0.06 (1.82)
  Week 48 (n=48) | -0.04 (2.81)

9. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Erosion of the Wrist and MCP Joints According to RAMRIS Score
Description: Erosion was evaluated at 15 sites in the wrist and 8 sites in the MCP joints. Bone erosion was scored on a scale of 0 to 10, where 0 represented no bone erosion and each 1-point increase reflected up to 10% increase in extent of erosion. Global RAMRIS scores were calculated as the sum of all joint sites for the wrist (range, 0 to 150) and MCP joints (range, 0 to 80). Aggregate wrist and MCP joint scores could range from 0 to 230 points. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in erosion.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
units on a scale
  Wrist Score, Baseline AV (n=56) | 7.32 (5.34)
  Wrist Score, Week 2 (n=46) | -0.24 (1.14)
  Wrist Score, Week 4 (n=50) | -0.16 (1.11)
  Wrist Score, Week 12 (n=51) | 0.08 (1.40)
  Wrist Score, Week 24 (n=50) | 0.28 (3.16)
  Wrist Score, Week 48 (n=47) | 0.34 (3.67)
  MCP Score, Baseline AV (n=54) | 4.26 (7.42)
  MCP Score, Week 2 (n=41) | -0.02 (0.88)
  MCP Score, Week 4 (n=47) | -0.04 (0.66)
  MCP Score, Week 12 (n=45) | 0.04 (1.19)
  MCP Score, Week 24 (n=46) | -0.07 (1.65)
  MCP Score, Week 48 (n=44) | 0.09 (1.18)
  Wrist and MCP Aggregate Score, Baseline AV (n=56) | 11.43 (9.98)
  Wrist and MCP Aggregate Score, Week 2 (n=46) | -0.39 (1.86)
  Wrist and MCP Aggregate Score, Week 4 (n=50) | -0.24 (1.55)
  Wrist and MCP Aggregate Score, Week 12 (n=51) | -0.41 (3.14)
  Wrist and MCP Aggregate Score, Week 24 (n=50) | -0.18 (4.77)
  Wrist and MCP Aggregate Score, Week 48 (n=47) | 0.36 (4.17)

10. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Number of Bones With Bone Marrow Edema in the Wrist and MCP Joints
Description: Edema was evaluated at 15 sites in the wrist and 8 sites in the MCP joints. Bone edema was scored on a scale of 0 to 3, where 0 represented no bone edema and each 1-point increase reflected one-third increase in extent of edema. The number of bones with edema was taken as the count of joints with a bone edema score greater than or equal to (≥) 1. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in edema.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bones with bone marrow edema
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
bones with bone marrow edema
  Baseline AV (n=56) | 7.91 (6.27)
  Week 2 (n=46) | -0.57 (3.46)
  Week 4 (n=50) | -0.78 (3.51)
  Week 12 (n=51) | -1.80 (3.98)
  Week 24 (n=50) | -2.56 (4.13)
  Week 48 (n=48) | -3.56 (5.07)

11. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Bone Marrow Edema of the Wrist and MCP Joints According to RAMRIS Score
Description: Edema was evaluated at 15 sites in the wrist and 8 sites in the MCP joints. Bone edema was scored on a scale of 0 to 3, where 0 represented no bone edema and each 1-point increase reflected one-third increase in extent of edema. Global RAMRIS scores were calculated as the sum of all joint sites for the wrist (range, 0 to 45) and MCP joints (range, 0 to 24). Aggregate wrist and MCP joint scores could range from 0 to 69 points. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in edema.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
units on a scale
  Wrist Score, Baseline AV (n=56) | 13.11 (12.88)
  Wrist Score, Week 2 (n=46) | -0.61 (6.23)
  Wrist Score, Week 4 (n=50) | -0.68 (5.87)
  Wrist Score, Week 12 (n=51) | -3.02 (8.55)
  Wrist Score, Week 24 (n=50) | -4.94 (10.80)
  Wrist Score, Week 48 (n=47) | -6.45 (11.90)
  MCP Score, Baseline AV (n=54) | 3.17 (4.64)
  MCP Score, Week 2 (n=41) | -0.32 (3.66)
  MCP Score, Week 4 (n=47) | -0.89 (4.17)
  MCP Score, Week 12 (n=45) | -1.47 (4.01)
  MCP Score, Week 24 (n=46) | -1.70 (3.35)
  MCP Score, Week 48 (n=44) | -1.98 (4.13)
  Wrist and MCP Aggregate Score, Baseline AV (n=56) | 16.16 (15.20)
  Wrist and MCP Aggregate Score, Week 2 (n=46) | -0.89 (7.71)
  Wrist and MCP Aggregate Score, Week 4 (n=50) | -1.52 (7.90)
  Wrist and MCP Aggregate Score, Week 12 (n=51) | -4.67 (9.29)
  Wrist and MCP Aggregate Score, Week 24 (n=50) | -6.70 (10.98)
  Wrist and MCP Aggregate Score, Week 48 (n=47) | -8.30 (13.06)

12. Secondary Outcome: Change From Baseline to Weeks 24 and 48 in Total Modified Sharp Score (TMSS), Erosion Score (ES), and Joint Space Narrowing Score (JSNS)
Description: The TMSS was calculated as the sum of ES and JSNS and ranged from 0 to 202. The ES was taken as the sum of joint scores collected for 14 joints in each hand (individually scored from 0 to 7) and ranged from 0 to 98 for both hands. The JSNS was the sum of joint scores collected for 13 joints in each hand (individually scored from 0 to 8) and ranged from 0 to 104 for both hands. Scores of 0 reflected no change, while higher scores reflected increased disease activity. Baseline AV and changes from Baseline to Weeks 24 and 48 were averaged among all participants, where negative changes indicated improvement in disease activity.
Time Frame: Baseline and Weeks 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 55
units on a scale
  TMSS, Baseline AV (n=55) | 18.25 (26.37)
  TMSS, Week 24 (n=46) | 0.41 (3.03)
  TMSS, Week 48 (n=47) | 1.46 (5.66)
  ES, Baseline AV (n=55) | 4.78 (11.85)
  ES, Week 24 (n=46) | 0.05 (0.60)
  ES, Week 48 (n=47) | 0.31 (1.07)
  JSNS, Baseline AV (n=55) | 13.46 (17.39)
  JSNS, Week 24 (n=46) | 0.36 (3.00)
  JSNS, Week 48 (n=47) | 1.15 (5.42)

13. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Ritchie Articular Index Score
Description: The Ritchie Articular Index was scored on a scale of 0 to 3, according to the grades of tenderness in each of 26 assessed joints. The total score was taken as the sum of joint scores and ranged from 0 to 78. Scores of 0 reflected no tenderness, while higher scores reflected increased tenderness. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in joint tenderness.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: ITT Population. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
units on a scale
  Baseline AV (n=58) | 16.69 (7.50)
  Week 2 (n=53) | -4.85 (5.37)
  Week 4 (n=54) | -7.06 (6.50)
  Week 12 (n=52) | -9.37 (6.65)
  Week 24 (n=53) | -11.60 (6.71)
  Week 48 (n=54) | -12.09 (6.95)

14. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Perceived Pain According to Visual Analog Scale (VAS) Score
Description: Perceived pain was assessed on a 0- to 100-millimeter (mm) VAS, where the distance from 0 mm represented the participant's self evaluation of pain (0 mm = no pain, 100 mm = maximum pain). Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated a decrease in perceived pain.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 54
mm
  Baseline AV (n=54) | 57.69 (24.07)
  Week 2 (n=50) | -18.56 (20.73)
  Week 4 (n=51) | -20.57 (22.44)
  Week 12 (n=52) | -32.75 (29.00)
  Week 24 (n=50) | -35.36 (24.62)
  Week 48 (n=50) | -39.44 (25.26)

15. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Perceived General Health According to VAS Score
Description: Global assessment of disease activity was performed using a 0- to 100-mm VAS, where the distance from 0 mm represented the investigator's evaluation or the participant's self evaluation of disease activity (0 mm = no disease activity, 100 mm = maximum disease activity). Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated improvement in disease activity.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 55
mm
  Participant Evaluation, Baseline AV (n=55) | 59.51 (23.32)
  Participant Evaluation, Week 2 (n=50) | -19.58 (20.75)
  Participant Evaluation, Week 4 (n=52) | -19.73 (23.46)
  Participant Evaluation, Week 12 (n=53) | -32.64 (28.59)
  Participant Evaluation, Week 24 (n=51) | -36.55 (23.84)
  Participant Evaluation, Week 48 (n=51) | -40.41 (25.69)
  Investigator Evaluation, Baseline AV (n=54) | 58.89 (16.26)
  Investigator Evaluation, Week 2 (n=47) | -19.21 (16.71)
  Investigator Evaluation, Week 4 (n=51) | -27.55 (20.49)
  Investigator Evaluation, Week 12 (n=51) | -37.61 (21.63)
  Investigator Evaluation, Week 24 (n=50) | -43.94 (19.55)
  Investigator Evaluation, Week 48 (n=50) | -44.72 (18.98)

16. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI assessed 20 items in eight functional activity domains including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item was scored on a scale of 0 to 3, where 0 represented activities performed without difficulty and 3 represented inability to perform activities alone. The total score was calculated as an average of all item scores, and thus also ranged from 0 to 3. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated an increase in ability to perform activities independently.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: ITT Population. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
units on a scale
  Baseline AV (n=58) | 1.33 (0.78)
  Week 2 (n=52) | -0.34 (0.51)
  Week 4 (n=53) | -0.35 (0.49)
  Week 12 (n=54) | -0.52 (0.68)
  Week 24 (n=53) | -0.61 (0.58)
  Week 48 (n=54) | -0.67 (0.61)

17. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Disease Activity Score of 28 Joints (DAS28) Score
Description: The DAS28 was derived from assessments of C-reactive protein (CRP), tender joint count (TJC), swollen joint count (SJC), and general health according to 100-mm VAS. DAS28 scores were calculated as [0.56 × square root of TJC] plus (+) [0.28 × square root of SJC] + [0.36 × natural log (CRP + 1)] + [0.014 × VAS] + 0.96. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. CRP was measured in milligrams per deciliter (mg/dL). DAS28 scores could range from 0 to 10, where higher scores represented higher disease activity. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: ITT Population. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
units on a scale
  Baseline AV (n=58) | 5.44 (0.90)
  Week 2 (n=50) | -1.22 (0.88)
  Week 4 (n=53) | -1.62 (1.05)
  Week 12 (n=53) | -2.29 (1.31)
  Week 24 (n=53) | -2.88 (1.17)
  Week 48 (n=53) | -3.07 (1.27)

18. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Vascular Endothelial Growth Factor (VEGF) Concentration
Description: Level of VEGF was measured in picograms per milliliter (pg/mL). Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 53
pg/mL
  Baseline AV (n=53) | 154.37 (130.97)
  Week 2 (n=45) | -53.06 (145.81)
  Week 4 (n=48) | -63.61 (121.55)
  Week 12 (n=47) | -36.33 (189.04)
  Week 24 (n=45) | -66.10 (139.38)
  Week 48 (n=45) | -29.35 (183.46)

19. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Erythrocyte Sedimentation Rate (ESR)
Description: ESR was measured in millimeters per hour (mm/h). Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
mm/h
  Baseline AV (n=56) | 37.39 (23.79)
  Week 2 (n=47) | -27.30 (20.08)
  Week 4 (n=52) | -27.63 (21.17)
  Week 12 (n=51) | -28.75 (23.00)
  Week 24 (n=50) | -30.58 (22.96)
  Week 48 (n=51) | -27.22 (21.79)

20. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in High-Sensitivity C-Reactive Protein (hsCRP) Concentration
Description: Level of hsCRP was measured in mg/dL. Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: ITT Population. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
mg/dL
  Baseline AV (n=58) | 14.43 (20.46)
  Week 2 (n=50) | -13.44 (21.56)
  Week 4 (n=53) | -11.96 (18.23)
  Week 12 (n=55) | -11.56 (22.51)
  Week 24 (n=53) | -13.43 (21.10)
  Week 48 (n=53) | -10.49 (12.31)

21. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Soluble Interleukin-6 Receptor (sIL6R) Level
Description: Level of sIL6R was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 45270.8 (19965.0)
  Week 2 (n=44) | 332597.2 (264433.0)
  Week 4 (n=50) | 303037.2 (253261.4)

22. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Messenger Ribonucleic Acid (mRNA) for Interleukin (IL)-17 (2^Delta Cycle Threshold [ΔCt]) Level
Description: Level of mRNA for IL-17 (2^ΔCt) was quantified by polymerase chain reaction (PCR). Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 2^ΔCt
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
2^ΔCt
  Baseline AV (n=51) | 0.0 (0.0)
  Week 2 (n=37) | 0.0 (0.0)
  Week 4 (n=44) | 0.0 (0.0)

23. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in mRNA for IL-23 Receptor (2^ΔCt) Level
Description: Level of mRNA for IL-23 receptor (2^ΔCt) was quantified by PCR. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 2^ΔCt
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 41
2^ΔCt
  Baseline AV (n=41) | 0.224 (0.415)
  Week 2 (n=31) | -0.007 (0.268)
  Week 4 (n=35) | 0.015 (0.495)

24. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in mRNA for RAR-Related Orphan Receptor (ROR)-γT (2^ΔCt) Level
Description: Level of ROR-γT (2^ΔCt) was quantified by PCR. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 2^ΔCt
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
2^ΔCt
  Baseline AV (n=51) | 0.083 (0.269)
  Week 2 (n=37) | -0.027 (0.259)
  Week 4 (n=44) | -0.004 (0.310)

25. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in mRNA for Forkhead Box Protein (FOXP) 3 (2^ΔCt) Level
Description: Level of mRNA for FOXP3 (2^ΔCt) was quantified by PCR. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 2^ΔCt
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
2^ΔCt
  Baseline AV (n=51) | 1.035 (2.509)
  Week 2 (n=37) | -0.315 (1.446)
  Week 4 (n=44) | -0.059 (1.615)

26. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Cluster of Differentiation (CD) 4-Positive Cells as a Percentage of Peripheral Blood Mononuclear Cells (PBMCs)
Description: The intensity of CD4-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
percentage of PBMCs
  Baseline AV (n=51) | 56.15 (12.63)
  Week 2 (n=29) | -1.47 (13.64)
  Week 4 (n=45) | 0.77 (8.97)

27. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD4 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD4-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
fluorescence intensity units
  Baseline AV (n=51) | 6970.94 (2725.05)
  Week 2 (n=29) | 464.04 (3341.91)
  Week 4 (n=45) | -1139.29 (3024.58)

28. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD25-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD25-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
percentage of PBMCs
  Baseline AV (n=51) | 7.27 (4.92)
  Week 2 (n=28) | -0.95 (6.54)
  Week 4 (n=45) | 0.04 (5.63)

29. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD25 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD25-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 51
fluorescence intensity units
  Baseline AV (n=51) | 2326.25 (923.68)
  Week 2 (n=28) | 74.76 (1850.13)
  Week 4 (n=45) | 162.27 (632.62)

30. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD45 "RO" Isoform (RO)-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD45RO-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 50
percentage of PBMCs
  Baseline AV (n=50) | 37.16 (11.50)
  Week 2 (n=23) | 1.77 (13.88)
  Week 4 (n=45) | 3.06 (11.65)

31. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD45RO Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD45RO-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 5138.47 (2184.11)
  Week 2 (n=22) | -1779.59 (2088.51)
  Week 4 (n=44) | -131.75 (1908.48)

32. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Cysteine-Cysteine Chemokine Receptor (CCR) 6-Positive Cells as a Percentage of PBMCs
Description: The intensity of CCR6-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
percentage of PBMCs
  Baseline AV (n=27) | 12.75 (6.40)
  Week 2 (n=19) | 2.34 (7.06)
  Week 4 (n=16) | 3.09 (6.76)

33. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CCR6 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CCR6-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
fluorescence intensity units
  Baseline AV (n=27) | 4651.85 (1211.33)
  Week 2 (n=19) | 291.63 (1820.02)
  Week 4 (n=16) | 376.56 (1306.58)

34. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CCR4-Positive Cells as a Percentage of PBMCs
Description: The intensity of CCR4-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
percentage of PBMCs
  Baseline AV (n=27) | 11.79 (5.45)
  Week 2 (n=19) | -1.64 (4.01)
  Week 4 (n=16) | 0.35 (3.11)

35. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CCR4 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CCR4-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
fluorescence intensity units
  Baseline AV (n=27) | 2534.67 (570.00)
  Week 2 (n=19) | 262.95 (755.79)
  Week 4 (n=16) | 273.19 (687.01)

36. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in IL-23 Receptor p19 Subunit (IL-23Rp19)-Positive Cells as a Percentage of PBMCs
Description: The intensity of IL-23Rp19-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
percentage of PBMCs
  Baseline AV (n=27) | 1.10 (1.19)
  Week 2 (n=19) | -0.32 (0.92)
  Week 4 (n=16) | -0.34 (0.49)

37. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in IL-23Rp19 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of IL-23Rp19-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
fluorescence intensity units
  Baseline AV (n=27) | 1416.30 (331.05)
  Week 2 (n=19) | 284.42 (1145.08)
  Week 4 (n=16) | 82.88 (552.61)

38. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Regulatory T (Treg) Cells as a Percentage of PBMCs
Description: The intensity of Treg cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 50
percentage of PBMCs
  Baseline AV (n=50) | 2.03 (1.02)
  Week 2 (n=39) | -0.07 (0.86)
  Week 4 (n=42) | 0.35 (1.41)

39. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Treg Cells as a Percentage of T Cells
Description: The intensity of Treg cell infiltration was expressed as the percentage of T cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of T cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 50
percentage of T cells
  Baseline AV (n=50) | 2.42 (1.18)
  Week 2 (n=39) | -0.19 (0.98)
  Week 4 (n=42) | 0.44 (1.80)

40. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Treg Cell Level
Description: The absolute number of Treg cells was expressed as cells per microliter (cells/mcL). Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
cells/mcL
  Baseline AV (n=49) | 34.51 (18.35)
  Week 2 (n=35) | 1.25 (13.75)
  Week 4 (n=42) | 6.30 (34.60)

41. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Helper T (Th) 17 Cells as a Percentage of PBMCs
Description: The intensity of Th17 cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
percentage of PBMCs
  Baseline AV (n=27) | 0.024 (0.036)
  Week 2 (n=18) | 0.006 (0.059)
  Week 4 (n=16) | -0.002 (0.064)

42. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Th17 Cells as a Percentage of T Cells
Description: The intensity of Th17 cell infiltration was expressed as the percentage of T cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of T cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
percentage of T cells
  Baseline AV (n=27) | 0.031 (0.049)
  Week 2 (n=18) | -0.003 (0.076)
  Week 4 (n=16) | -0.007 (0.027)

43. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Th17 Cell Level
Description: The absolute number of Th17 cells was expressed as cells/mcL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 27
cells/mcL
  Baseline AV (n=27) | 0.295 (0.368)
  Week 2 (n=18) | 0.050 (0.344)
  Week 4 (n=17) | -0.068 (0.288)

44. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD19-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD19-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 8.40 (4.68)
  Week 2 (n=1) | -4.80 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.12 (6.39)

45. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD19 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD19-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 19268.58 (5482.10)
  Week 2 (n=1) | -3656.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 251.34 (5251.35)

46. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD24-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD24-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 8.02 (4.64)
  Week 2 (n=1) | -4.90 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.73 (6.21)

47. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD24 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD24-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 3133.63 (1652.36)
  Week 2 (n=1) | 1015.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 436.05 (1827.22)

48. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD27-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD27-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 57.51 (16.48)
  Week 2 (n=1) | -12.40 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 1.44 (12.22)

49. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD27 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD27-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 1288.10 (302.90)
  Week 2 (n=1) | -349.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -53.98 (390.89)

50. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD38-Positive Cells as a Percentage of PBMCs
Description: The intensity of CD38-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 49.51 (11.51)
  Week 2 (n=1) | -4.30 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.78 (10.87)

51. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in CD38 Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of CD38-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 5746.98 (2082.63)
  Week 2 (n=1) | -193.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 162.66 (1602.09)

52. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Immunoglobulin (Ig) M-Positive Cells as a Percentage of PBMCs
Description: The intensity of IgM-positive cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 17.06 (14.50)
  Week 2 (n=1) | -3.60 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 1.19 (11.61)

53. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in IgM Mean Intensity of Fluorescence
Description: The mean fluorescence intensity of IgM-positive cells was measured by flow cytometry. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fluorescence intensity units
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
fluorescence intensity units
  Baseline AV (n=49) | 15545.94 (7231.80)
  Week 2 (n=1) | -10381.0 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -56.45 (5681.03)

54. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Mature B Cells as a Percentage of PBMCs
Description: The intensity of mature B cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 4.72 (3.56)
  Week 2 (n=1) | -3.40 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.35 (4.24)

55. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Mature B Cells as a Percentage of B Cells
Description: The intensity of mature B cell infiltration was expressed as the percentage of B cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of B cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of B cells
  Baseline AV (n=49) | 48.58 (14.72)
  Week 2 (n=1) | -9.40 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.11 (13.79)

56. Secondary Outcome: Change From Baseline to Week 4 in Mature B Cell Level
Description: The absolute number of mature B cells was expressed as cells/mcL. Baseline AV and change from Baseline to Week 4 were averaged among all participants.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 47
cells/mcL
  Baseline AV (n=47) | 78.27 (73.37)
  Week 4 (n=42) | 2.29 (74.72)

57. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Memory B Cells as a Percentage of PBMCs
Description: The intensity of memory B cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 1.49 (1.56)
  Week 2 (n=1) | -0.90 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 0.13 (1.28)

58. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Memory B Cells as a Percentage of B Cells
Description: The intensity of memory B cell infiltration was expressed as the percentage of B cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of B cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of B cells
  Baseline AV (n=49) | 18.95 (13.36)
  Week 2 (n=1) | 4.30 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | 0.62 (10.87)

59. Secondary Outcome: Change From Baseline to Week 4 in Memory B Cell Level
Description: The absolute number of memory B cells was expressed as cells/mcL. Baseline AV and change from Baseline to Week 4 were averaged among all participants.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 47
cells/mcL
  Baseline AV (n=47) | 29.29 (40.81)
  Week 4 (n=42) | 2.85 (37.60)

60. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Transitional B Cells as a Percentage of PBMCs
Description: The intensity of transitional B cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 0.58 (1.12)
  Week 2 (n=1) | 0.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.22 (1.21)

61. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Transitional B Cells as a Percentage of B Cells
Description: The intensity of transitional B cell infiltration was expressed as the percentage of B cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of B cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of B cells
  Baseline AV (n=49) | 5.26 (5.61)
  Week 2 (n=1) | 5.80 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -1.09 (4.54)

62. Secondary Outcome: Change From Baseline to Week 4 in Transitional B Cell Level
Description: The absolute number of transitional B cells was expressed as cells/mcL. Baseline AV and change from Baseline to Week 4 were averaged among all participants.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 47
cells/mcL
  Baseline AV (n=47) | 6.70 (7.79)
  Week 4 (n=42) | -0.62 (7.51)

63. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Plasma B Cells as a Percentage of PBMCs
Description: The intensity of plasma B cell infiltration was expressed as the percentage of PBMCs. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PBMCs
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of PBMCs
  Baseline AV (n=49) | 0.22 (0.57)
  Week 2 (n=1) | 0.00 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.08 (0.60)

64. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Plasma B Cells as a Percentage of B Cells
Description: The intensity of plasma B cell infiltration was expressed as the percentage of B cells. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of B cells
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
percentage of B cells
  Baseline AV (n=49) | 1.52 (4.54)
  Week 2 (n=1) | -0.20 (NA) — Standard deviation could not be calculated because the analysis only included 1 participant.
  Week 4 (n=44) | -0.06 (5.77)

65. Secondary Outcome: Change From Baseline to Week 4 in Plasma B Cell Level
Description: The absolute number of plasma B cells was expressed as cells/mcL. Baseline AV and change from Baseline to Week 4 were averaged among all participants.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 47
cells/mcL
  Baseline AV (n=47) | 3.13 (6.50)
  Week 4 (n=42) | -1.11 (6.31)

66. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Th17 Cysteine-Cysteine Chemokine Ligand (CCL) 20 Level
Description: Level of Th17CCL20 was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 35.03 (69.50)
  Week 2 (n=46) | 2.57 (20.72)
  Week 4 (n=52) | -2.65 (23.18)

67. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Th17CCL17 Level
Description: as for outcome 66
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
pg/mL
  Baseline AV (n=56) | 456.02 (404.17)
  Week 2 (n=45) | 119.58 (453.39)
  Week 4 (n=51) | 75.84 (333.43)

68. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in B Cell-Attracting Chemokine (BCA) Level
Description: Level of BCA was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 56
pg/mL
  Baseline AV (n=56) | 122.28 (87.48)
  Week 2 (n=45) | -21.37 (70.40)
  Week 4 (n=51) | -18.26 (103.62)

69. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Stromal Cell-Derived Factor (SDF) 1 Level
Description: Level of SDF1 was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 2151.47 (1133.79)
  Week 2 (n=46) | -1.85 (343.10)
  Week 4 (n=52) | -26.46 (390.80)

70. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in B Cell-Activating Factor (BAFF) Level
Description: Level of BAFF was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 802.98 (317.98)
  Week 2 (n=45) | 28.04 (217.89)
  Week 4 (n=52) | 36.17 (223.64)

71. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in A Proliferation-Inducing Ligand (APRIL) Level
Description: Level of APRIL was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 6807.49 (11178.42)
  Week 2 (n=45) | -816.13 (4036.61)
  Week 4 (n=51) | 7.82 (3843.69)

72. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Tumor Necrosis Factor (TNF)-α Level
Description: Level of TNF-α was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 55
pg/mL
  Baseline AV (n=55) | 2.285 (4.234)
  Week 2 (n=42) | 0.077 (1.228)
  Week 4 (n=46) | 0.254 (0.978)

73. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in IL-1β Level
Description: Level of IL-1β was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 37
pg/mL
  Baseline AV (n=37) | 0.699 (0.692)
  Week 2 (n=27) | -0.160 (0.598)
  Week 4 (n=31) | -0.243 (0.620)

74. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in IL-17 Level
Description: Level of IL-17 was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 15.00 (0.00)
  Week 2 (n=47) | 0.00 (0.00)
  Week 4 (n=52) | 0.00 (0.00)

75. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Monocyte Chemoattractant Protein (MCaP)-1 Level
Description: Level of MCaP-1 was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 343.86 (283.29)
  Week 2 (n=47) | 22.70 (143.82)
  Week 4 (n=51) | -33.20 (133.52)

76. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Osteocalcin Level
Description: Level of osteocalcin was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 14069.60 (8770.17)
  Week 2 (n=47) | -616.34 (6899.51)
  Week 4 (n=52) | -99.00 (6938.56)

77. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Type I Collagen N-Propeptide Level
Description: Level of Type I collagen N-propeptide was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 7731.89 (4625.23)
  Week 2 (n=46) | 842.65 (4318.91)
  Week 4 (n=51) | -576.49 (4108.27)

78. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in C-Terminal Telopeptide (CTX)-1 Level
Description: Level of CTX-1 was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 487.28 (248.61)
  Week 2 (n=48) | 43.33 (193.11)
  Week 4 (n=50) | 48.80 (233.25)

79. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Type I Collagen C-Terminal Telopeptide (ICTP) Level
Description: Level of ICTP was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 6381.12 (2456.54)
  Week 2 (n=48) | 306.60 (1568.45)
  Week 4 (n=51) | 193.25 (1657.43)

80. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Type II Collagen N-Propeptide (PIIANP) Level
Description: Level of PIIANP was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 1329158 (908163.5)
  Week 2 (n=47) | -37518.8 (1008994)
  Week 4 (n=51) | -69799.1 (673406.7)

81. Secondary Outcome: Change From Baseline to Weeks 2 and 4 in Type II Collagen Helical Peptide (HELIX-II) Level
Description: Level of HELIX-II was measured in pg/mL. Baseline AV and changes from Baseline to Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 2521.12 (1960.76)
  Week 2 (n=48) | 126.02 (1480.97)
  Week 4 (n=51) | -78.29 (1586.43)

82. Secondary Outcome: Change From Baseline to Weeks 2, 4, 12, 24, and 48 in Hemoglobin (Hb) Concentration
Description: Level of Hb was measured in grams per liter (g/L). Baseline AV and changes from Baseline to Weeks 2, 4, 12, 24, and 48 were averaged among all participants.
Time Frame: Baseline and Weeks 2, 4, 12, 24, 48
Population: ITT Population. The number of participants who contributed to the analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 58
g/L
  Baseline AV (n=58) | 128.28 (12.10)
  Week 2 (n=50) | 3.86 (5.87)
  Week 4 (n=54) | 2.09 (5.35)
  Week 12 (n=55) | 4.31 (9.13)
  Week 24 (n=53) | 6.23 (8.99)
  Week 48 (n=53) | 7.17 (8.28)

83. Secondary Outcome: Change From Baseline to Day 2 and Weeks 2 and 4 in Soluble Transferrin Receptor (STR) Concentration
Description: Level of STR was measured in pg/mL. Baseline AV and changes from Baseline to Day 2 and Weeks 2 and 4 were averaged among all participants.
Time Frame: Baseline; Day 2; and Weeks 2, 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 57
pg/mL
  Baseline AV (n=57) | 4536413 (1336641)
  Day 2 (n=10) | -83532.0 (446321.3)
  Week 2 (n=46) | 15712.17 (821775.0)
  Week 4 (n=52) | -89722.7 (959232.1)

84. Secondary Outcome: Change From Baseline to Week 48 in Initial Rate of Enhancement (IRE) by DYNAMIKA Software Analysis
Description: IRE was approximated by parametric mapping via DYNAMIKA software and expressed as change in relative signal intensity per second (ΔI/sec). The mean of three different slices was used in the determination of IRE. Each slice consisted of a two-dimensional (2D) sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ΔI/sec
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
ΔI/sec
  Baseline AV (n=49) | 0.00503 (0.00371)
  Week 48 (n=32) | -0.00246 (0.00363)

85. Secondary Outcome: Change From Baseline to Week 48 in Maximum Enhancement (ME) by DYNAMIKA Software Analysis
Description: ME was approximated by parametric mapping via DYNAMIKA software and expressed as ratio of signal enhancement before and after contrast injection. The mean of three different slices was used in the determination of ME. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
ratio
  Baseline AV (n=49) | 1.606 (0.422)
  Week 48 (n=32) | -0.177 (0.416)

86. Secondary Outcome: Change From Baseline to Week 48 in Number of Enhancing Voxels (Ntotal) by DYNAMIKA Software Analysis
Description: Ntotal was approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Ntotal. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: enhancing voxels
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 48
enhancing voxels
  Baseline AV (n=48) | 3155.69 (1677.22)
  Week 48 (n=31) | -974.16 (1606.14)

87. Secondary Outcome: Change From Baseline to Week 48 in Number of Persistent Enhancing Voxels (Npersistent) by DYNAMIKA Software Analysis
Description: Npersistent was approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Npersistent. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: persistent enhancing voxels
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
persistent enhancing voxels
  Baseline AV (n=49) | 182.04 (157.15)
  Week 48 (n=32) | -0.53 (219.74)

88. Secondary Outcome: Change From Baseline to Week 48 in Number of Plateau Enhancing Voxels (Nplateau) by DYNAMIKA Software Analysis
Description: Nplateau was approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Nplateau. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: plateau enhancing voxels
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
plateau enhancing voxels
  Baseline AV (n=49) | 1839.63 (994.07)
  Week 48 (n=32) | -635.72 (1019.13)

89. Secondary Outcome: Change From Baseline to Week 48 in Number of Washout Enhancing Voxels (Nwashout) by DYNAMIKA Software Analysis
Description: Nwashout was approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Nwashout. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: washout enhancing voxels
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 49
washout enhancing voxels
  Baseline AV (n=49) | 1167.16 (783.19)
  Week 48 (n=32) | -358.25 (798.88)

90. Secondary Outcome: Change From Baseline to Week 48 in Ntotal×IRE by DYNAMIKA Software Analysis
Description: Ntotal and IRE were approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Ntotal. The mean of three different slices was used in the determination of IRE. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Function of Ntotal×IRE was expressed as voxels times change in relative intensity per second (v*ΔI/sec). Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: v*ΔI/sec
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 48
v*ΔI/sec
  Baseline AV (n=48) | 6.01 (5.93)
  Week 48 (n=31) | -4.84 (6.13)

91. Secondary Outcome: Change From Baseline to Week 48 in Ntotal×ME by DYNAMIKA Software Analysis
Description: Ntotal and ME were approximated using DYNAMIKA software. The sum of three different slices was used in the determination of Ntotal. The mean of three different slices was used in the determination of ME. Each slice consisted of a 2D sequence of images acquired from the same physical location at different time instances. Function of NtotalME was expressed as voxels times ratio of signal intensity before and after contrast injection (v*ratio). Baseline AV and change from Baseline to Week 48 were averaged among all participants.
Time Frame: Baseline and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: v*ratio
Arm/Group | Tocilizumab in Active RA
Number analyzed (Participants) | 48
v*ratio
  Baseline AV (n=48) | 1882.40 (1267.48)
  Week 48 (n=31) | -793.59 (1168.57)

ADVERSE EVENTS:
Time Frame: Baseline to Week 48
Description: Safety Population (same as ITT Population): All enrolled participants who received at least one dose of study drug.
Arm/Group | Tocilizumab in Active RA
Serious Adverse Events (participants affected / at risk) | 5/58
Other Adverse Events (participants affected / at risk) | 50/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab in Active RA (N=58)
Tachycardia (Cardiac disorders) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal colic (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab in Active RA (N=58)
Anaemia (Blood and lymphatic system disorders) | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 8
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Eyelid oedema (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dysentery (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Oropharyngeal pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
Face oedema (General disorders) | 1
Hyperpyrexia (General disorders) | 1
Pyrexia (General disorders) | 3
Swelling (General disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 5
Cystitis (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Labyrinthitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 7
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Eye injury (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 3
Blood phosphorus increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 8
Eosinophil count increased (Investigations) | 2
Lipids increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Transaminases increased (Investigations) | 5
White blood cell count decreased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Syncope (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Tachycardia (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.